CLINICAL TRIAL: NCT06618573
Title: Study on the Safety of Administering Isoniazid to Systemic Lupus Erythematosus Patients to Prevent Tuberculosis
Brief Title: Safety of Administering Isoniazid to SLE Patients to Prevent TB
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IPD-202402.01
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Tuberculosis; Systemic Lupus Erythematosus
Keywords: Tuberculosis; Systemic Lupus Erythematosus
MeSH Terms: conditions — Tuberculosis; Lupus Erythematosus, Systemic | interventions — Isoniazid; Pyridoxine

STUDY DESIGN:
Intervention Model Description: SLE patient at the Hasan Sadikin Rheumatology Outpatient Clinic and registered as Lupus Registry study participants with remission or mild SLE disease activity. Subjects fulfilled inclusion criteria will be randomly divided into two groups: treatment group receiving INH 5 mg/kg/day (maximum 300 mg/day) with pyridoxine 10 mg/day and control group receiving placebo.
  Monitor ALT/AST and SLE disease activity after two weeks, continued monthly for the first three months (1st, 2nd, 3rd) then every three months for up to a year (6th, 9th, 12th months). Routine SLE medication is continued and routinely recorded at every visit.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): SLE patient at the Hasan Sadikin Rheumatology Outpatient Clinic and registered as Lupus Registry with remission or mild SLE disease activity. The diagnosis of SLE is based on ACR 1997 criteria or SLE SLICC 2012 criteria. Screening will include history review, physical examinations, chest X-Ray, laboratory test such as CBC, ALT/AST, HbsAg, total anti-HCV, complement (C3), dsDNA, creatinine serum, urinalysis (proteinuria, ACR, RBC, WBC, casts), IGRA, to assess if any subject has no active TB and no chronic liver disease.
  Treatment group receiving Isoniazid 5 mg/kg/day (maximum 300 mg/day) with pyridoxine 10 mg/day.
  Monitor ALT/AST and SLE disease activity after two weeks, continued monthly for the first three months (1st, 2nd, 3rd) then every three months for up to a year (6th, 9th, 12th months). Routine SLE medication is continued and routinely recorded at every visit.
  Interventions: Drug: Isoniazid/Pyridoxine
- Control Group (Placebo Comparator): SLE patient at the Hasan Sadikin Rheumatology Outpatient Clinic and registered as Lupus Registry with remission or mild SLE disease activity. The diagnosis of SLE is based on ACR 1997 criteria or SLE SLICC 2012 criteria. Screening will include history review, physical examinations, chest X-ray, laboratory test such as CBC, ALT/AST, HbsAg, total anti-HCV, complement (C3), dsDNA, creatinine serum, urinalysis (proteinuria, ACR, RBC, WBC, casts) IGRA, to assess if any subject has no active TB and no chronic liver disease.
  Control group receiving placebo.
  Monitor ALT/AST and SLE disease activity after two weeks, continued monthly for the first three months (1st, 2nd, 3rd) then every three months for up to a year (6th, 9th, 12th months). Routine SLE medication is continued and routinely recorded at every visit.
  Interventions: Drug: Saccharum Lactis

INTERVENTIONS:
Drug: Isoniazid/Pyridoxine — Treatment group received isoniazid 300mg and pyridoxine 10mg/day
  Arms: Treatment Group
Drug: Saccharum Lactis — Control group received placebo
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
Systemic Lupus Erythematosus (SLE) is a prototypical systemic autoimmune disease characterized by heterogeneity, multisystem involvement, and production of multiple autoantibodies. Clinical features can vary, from mild skin and joint involvement to severe and life-threatening conditions.

Patients with lupus are more susceptible to infections, in addition to being immunocompromised, and due to the administration of corticosteroid and cytotoxic drugs. The presence of these infections is a cause of death in lupus disease in addition to the activity of the disease itself, especially in Asia-Pacific countries. One infection that often occurs in lupus is Tuberculosis (TB).

Efforts have been made to prevent TB infection in vulnerable populations, including isoniazid (INH) prophylaxis. In 2010, World Heatlh Organization issued guidelines for HIV patients to receive INH prophylaxis to prevent TB infection. The implementation of Isoniazid Preventive Therapy (IPT) is quite cheap using INH with mild side effects.18 A meta-analysis study of INH prophylaxis in patients with HIV found that the efficacy of this prophylaxis significantly reduced TB incidence by 35% with an RR of 0.65%. In addition, INH was found to be safe, with no significant increase in drug reactions, according to a meta-analysis of prophylaxis studies in HIV patients.

However, there is no guideline for INH prophylaxis for SLE patients, as there is for HIV patients, due to lack of data on this issue.

Studies on the effectiveness of INH prophylaxis on the prevention of TB infection for SLE patients should be conducted, but before that, studies on the safety of INH therapy in SLE patients should be conducted.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a prototypical systemic autoimmune disease characterized by heterogeneity, multisystem involvement, and production of multiple autoantibodies. Clinical features can vary, from mild skin and joint involvement to severe and life-threatening conditions. The course of lupus is highly variable in the form of relapses and remissions, with mild and severe forms that can be life-threatening. Treatments for SLE includes steroids and immunosuppressants to control disease activity.

Patients with lupus are more susceptible to infections, in addition to being immunocompromised, and due to the administration of corticosteroid and cytotoxic drugs. The presence of these infections is a cause of death in lupus disease in addition to the activity of the disease itself, especially in Asia-Pacific countries. One infection that often occurs in lupus is Tuberculosis (TB).

Tuberculosis is still a problem especially in the Asian region, and Indonesia ranks 2nd with the most cases after India according to World Health Organization in 2019. TB infection is found in 10-11.4% of SLE patients in Asia. The incidence of TB in SLE is reported to range from 150/100,000 patients per year in Turkey to 2,450/100,000 patients per year in India. The annual risk of TB in SLE patients is higher than the normal population. Registry data at Hasan Sadikin Hospital Bandung showed that 11.4% or 93 out of 813 SLE patients were infected with TB after being diagnosed with SLE.

Risk factors for increased TB infection in SLE patients, in addition to SLE disease activity itself (SLEDAI score >12), renal involvement, lymphopenia, and cumulative dose of steroids used by the patient, are also due to long duration of illness and previous history of TB.

Tuberculosis is also one of the infections that cause death in SLE patients. Mortality from TB in Asian countries ranged from 5-31%. A study in the Philippines found that 14.8% of SLE patients with TB died, those who died had disseminated TB or miliary TB.

Efforts have been made to prevent TB infection in vulnerable populations, including isoniazid (INH) prophylaxis. In 2010, World Health Organization issued guidelines for HIV patients to receive INH prophylaxis to prevent TB infection. The implementation of Isoniazid Preventive Therapy (IPT) is quite cheap using INH with mild side effects. A meta-analysis study of INH prophylaxis in patients with HIV found that the efficacy of this prophylaxis significantly reduced TB incidence by 35% with an RR of 0.65%. In addition, INH was found to be safe, with no significant increase in drug reactions, according to a meta-analysis of prophylaxis studies in HIV patients.

The role of isoniazid prophylaxis for TB prevention in patients with SLE is controversial. To date, there is no consensus on prophylaxis against TB in SLE patients.

Research on this prophylaxis has been presented in an Indian study by Gaitonde et al. They found an 82% reduction in TB incidence in SLE patients with prophylactic INH at 5 mg/kg/day, with a maximum dose of 300 mg/day plus 10 mg pyridoxine (Vitamin B6) for 1 year, and no significant liver toxicity due to this drug. However, a retrospective study conducted in Hong Kong found no significant difference in TB reactivation between those who received INH compared to those who did not receive INH, while patients who received INH were reported to have more relapses of their lupus. Similarly, a retrospective study in Korea found no significant difference in patients with lupus nephritis.

The high incidence of TB in SLE patients, especially in endemic areas such as Indonesia, makes TB prevention an important endeavour. However, there is no guideline for INH prophylaxis for SLE patients, as there is for HIV patients, due to lack of data on this issue.

Studies on the effectiveness of INH prophylaxis on the prevention of TB for SLE patients should be conducted, but before that, studies on the safety of INH therapy in SLE patients should be conducted.

This study was a cohort study, with the following research design:

* LES patients attending the rheumatology clinic of RSHS and enrolled as Lupus Registry study participants, with remission or mild SLE disease activity
* Screening for TB and impaired liver function (Informed Consent, history review, physical examination, laboratory examination, Chest X-Ray) -> Exclude if have condition: Impaired liver function, including hepatitis B/C positivity, history of allergy to INH, pregnancy, malignancy
* SLE patients who fulfil the inclusion criteria divided into two groups: Received INH 300 mg/day and Pyridoxine 10 mg/day for nine months or placebo.
* Routine SLE medication continued and routinely recorded at each visit.
* Monitor SGOT/SGPT and SLE disease activity after two weeks, continuing monthly in the first three months (months 1/2 1, 2, 3) then every three months until one year (months 6, 9, 12).

Inclusion Criteria:

* SLE patients with conditions of:
* No signs and symptoms of active TB,
* Not under TB treatment,
* No History of TB, malignancy, HIV, liver function test abnormality
* Not in pregnancy/lactation,
* No other active infections
* Remission or low to moderate disease activity state,
* Consented to join the study completely.

Exclusion Criteria:

* SLE patients with conditions of:
* History of allergy to Isoniazid,
* Chronic liver disease, including chronic hepatitis B or C virus,
* Malignancy,
* Pregnancy.

The patients included were patients who had been diagnosed with SLE and were registered in Lupus Registry.

The study was explained and informed consent was obtained. After the patient agreed and signed Informed Consent, screening was conducted to ensure that there was no active TB, impaired liver function (SGOT/SGPT), positive Hepatitis B (HBsAg) and/or Hepatitis C (total Anti HCV), history of Isoniazid (INH) allergy, history of malignancy, and pregnancy. If any of these conditions exist, the subject will be excluded.

Eligible subjects were randomly grouped into two groups: those receiving INH 5 mg/kg/day (maximum 300 mg/day) & Pyridoxine (Vitamin B6) 10 mg/day, or placebo. Other routine SLE medications were continued.

Sample calculations were carried out based on INH prophylaxis studies conducted in HIV patients, obtaining a risk of drug reaction events of RR 1.2, so that with a confidence level of 95% and 80% power and an effect size of 0.5, the sample size for each group was 27 people, plus 10% to 30 people. So that the total number of patients involved is 60 people divided into 2 groups.

This study was to assess the safety of INH drug administration to lupus patients assessed by the increase in SGPT and SGOT that occurred and their lupus disease activity (using the SLEDAI score) measured at month 1/2 (second week), 1, 2, 3, 6, 9 and 12. The statistical test used was a T-test comparing two groups.

The study was conducted at Dr. Hasan Sadikin Hospital, Bandung. The study was conducted from August 2022 to December 2024.

ELIGIBILITY:
Inclusion Criteria:

SLE patients with conditions of :

* No signs and symptoms of active TB
* Not under TB treatment
* No History of TB, malignancy, HIV, liver function test abnormality
* Not in pregnancy/lactation
* No other active infections
* Remission or low to moderate disease activity state
* Consented to join the study completely

Exclusion Criteria:

SLE patients with conditions of :

* History of allergy to Isoniazid
* Chronic liver disease, including chronic hepatitis B or C virus
* Malignancy
* Pregnancy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Drug Induce Hepatitis | week 2, months 1, 2, 3, 6, 9, 12
  Change in more than twice the upper limit of normal SGOT/SGPT values and improvement after drug discontinuation
SLE disease activity | month 1, 2, 3, 6, 9, 12
  Based on Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score. The higher the score, the worse. SLEDAI score increase in more than 3=flare

CONTACTS AND LOCATIONS:
Overall Officials: Laniyati Hamijoyo, MD, PhD, Principal Investigator — Universitas Padjadjaran
Locations (1):
- Rumah Sakit Dr Hasan Sadikin, Universitas Padjadjaran, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamijoyo L, Candrianita S, Rahmadi AR, Dewi S, Darmawan G, Suryajaya BS, Rainy NR, Hidayat II, Moenardi VN, Wachjudi RG. The clinical characteristics of systemic lupus erythematosus patients in Indonesia: a cohort registry from an Indonesia-based tertiary referral hospital. Lupus. 2019 Nov;28(13):1604-1609. doi: 10.1177/0961203319878499. Epub 2019 Sep 29. PMID 31566078
- [Background] Koesoemadinata RC, McAllister SM, Soetedjo NNM, Febni Ratnaningsih D, Ruslami R, Kerry S, Verrall AJ, Apriani L, van Crevel R, Alisjahbana B, Hill PC. Latent TB infection and pulmonary TB disease among patients with diabetes mellitus in Bandung, Indonesia. Trans R Soc Trop Med Hyg. 2017 Feb 1;111(2):81-89. doi: 10.1093/trstmh/trx015. PMID 28419376
- [Background] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Background] Yu YC, Mao YM, Chen CW, Chen JJ, Chen J, Cong WM, Ding Y, Duan ZP, Fu QC, Guo XY, Hu P, Hu XQ, Jia JD, Lai RT, Li DL, Liu YX, Lu LG, Ma SW, Ma X, Nan YM, Ren H, Shen T, Wang H, Wang JY, Wang TL, Wang XJ, Wei L, Xie Q, Xie W, Yang CQ, Yang DL, Yu YY, Zeng MD, Zhang L, Zhao XY, Zhuang H; Drug-induced Liver Injury (DILI) Study Group; Chinese Society of Hepatology (CSH); Chinese Medical Association (CMA). CSH guidelines for the diagnosis and treatment of drug-induced liver injury. Hepatol Int. 2017 May;11(3):221-241. doi: 10.1007/s12072-017-9793-2. Epub 2017 Apr 12. PMID 28405790
- [Background] Hochberg MC. Updating the American College of Rheumatology revised criteria for the classification of systemic lupus erythematosus. Arthritis Rheum. 1997 Sep;40(9):1725. doi: 10.1002/art.1780400928. No abstract available. PMID 9324032
- [Background] Victorio-Navarra ST, Dy EE, Arroyo CG, Torralba TP. Tuberculosis among Filipino patients with systemic lupus erythematosus. Semin Arthritis Rheum. 1996 Dec;26(3):628-34. doi: 10.1016/s0049-0172(96)80013-8. PMID 8989807
- [Background] Pattanaik SS, Muhammed H, Chatterjee R, Naveen R, Lawrence A, Agarwal V, Misra DP, Gupta L, Misra R, Aggarwal A. In-hospital mortality and its predictors in a cohort of SLE from Northern India. Lupus. 2020 Dec;29(14):1971-1977. doi: 10.1177/0961203320961474. Epub 2020 Sep 30. PMID 32998621
- [Background] Lao M, Chen D, Wu X, Chen H, Qiu Q, Yang X, Zhan Z. Active tuberculosis in patients with systemic lupus erythematosus from Southern China: a retrospective study. Clin Rheumatol. 2019 Feb;38(2):535-543. doi: 10.1007/s10067-018-4303-z. Epub 2018 Sep 23. PMID 30244432
- [Background] Mok MY, Lo Y, Chan TM, Wong WS, Lau CS. Tuberculosis in systemic lupus erythematosus in an endemic area and the role of isoniazid prophylaxis during corticosteroid therapy. J Rheumatol. 2005 Apr;32(4):609-15. PMID 15801014
- [Background] Tam LS, Li EK, Wong SM, Szeto CC. Risk factors and clinical features for tuberculosis among patients with systemic lupus erythematosus in Hong Kong. Scand J Rheumatol. 2002;31(5):296-300. doi: 10.1080/030097402760375205. PMID 12455821
- [Background] Ahmmed MF, Islam MN, Ferdous S, Azad AK, Ferdous N. Tuberculosis in Systemic Lupus Erythematosus Patients. Mymensingh Med J. 2019 Oct;28(4):797-807. PMID 31599243
- [Background] Jakes RW, Bae SC, Louthrenoo W, Mok CC, Navarra SV, Kwon N. Systematic review of the epidemiology of systemic lupus erythematosus in the Asia-Pacific region: prevalence, incidence, clinical features, and mortality. Arthritis Care Res (Hoboken). 2012 Feb;64(2):159-68. doi: 10.1002/acr.20683. PMID 22052624
- [Background] Lisnevskaia L, Murphy G, Isenberg D. Systemic lupus erythematosus. Lancet. 2014 Nov 22;384(9957):1878-1888. doi: 10.1016/S0140-6736(14)60128-8. Epub 2014 May 31. PMID 24881804
- [Background] Iliopoulos AG, Tsokos GC. Immunopathogenesis and spectrum of infections in systemic lupus erythematosus. Semin Arthritis Rheum. 1996 Apr;25(5):318-36. doi: 10.1016/s0049-0172(96)80018-7. PMID 8778988
- [Background] Yun JE, Lee SW, Kim TH, Jun JB, Jung S, Bae SC, Kim TY, Yoo DH. The incidence and clinical characteristics of Mycobacterium tuberculosis infection among systemic lupus erythematosus and rheumatoid arthritis patients in Korea. Clin Exp Rheumatol. 2002 Mar-Apr;20(2):127-32. PMID 12051389
- [Background] Erdozain JG, Ruiz-Irastorza G, Egurbide MV, Martinez-Berriotxoa A, Aguirre C. High risk of tuberculosis in systemic lupus erythematosus? Lupus. 2006;15(4):232-5. doi: 10.1191/0961203306lu2289xx. PMID 16686263
- [Background] Sayarlioglu M, Inanc M, Kamali S, Cefle A, Karaman O, Gul A, Ocal L, Aral O, Konice M. Tuberculosis in Turkish patients with systemic lupus erythematosus: increased frequency of extrapulmonary localization. Lupus. 2004;13(4):274-8. doi: 10.1191/0961203303lu529xx. PMID 15176665
- [Background] Shyam C, Malaviya AN. Infection-related morbidity in systemic lupus erythematosus: a clinico-epidemiological study from northern India. Rheumatol Int. 1996;16(1):1-3. doi: 10.1007/BF01419946. PMID 8783414
- [Background] Bharath G, Kumar P, Makkar N, Singla P, Soneja M, Biswas A, Wig N. Mortality in systemic lupus erythematosus at a teaching hospital in India: A 5-year retrospective study. J Family Med Prim Care. 2019 Jul;8(7):2511-2515. doi: 10.4103/jfmpc.jfmpc_362_19. PMID 31463286
- [Background] Ayele HT, Mourik MS, Debray TP, Bonten MJ. Isoniazid Prophylactic Therapy for the Prevention of Tuberculosis in HIV Infected Adults: A Systematic Review and Meta-Analysis of Randomized Trials. PLoS One. 2015 Nov 9;10(11):e0142290. doi: 10.1371/journal.pone.0142290. eCollection 2015. PMID 26551023
- [Background] Gaitonde S, Pathan E, Sule A, Mittal G, Joshi VR. Efficacy of isoniazid prophylaxis in patients with systemic lupus erythematosus receiving long term steroid treatment. Ann Rheum Dis. 2002 Mar;61(3):251-3. doi: 10.1136/ard.61.3.251. PMID 11830432
- [Background] Polachek A, Gladman DD, Su J, Urowitz MB. Defining Low Disease Activity in Systemic Lupus Erythematosus. Arthritis Care Res (Hoboken). 2017 Jul;69(7):997-1003. doi: 10.1002/acr.23109. PMID 27696791
- [Background] Mikdashi J, Nived O. Measuring disease activity in adults with systemic lupus erythematosus: the challenges of administrative burden and responsiveness to patient concerns in clinical research. Arthritis Res Ther. 2015 Jul 20;17(1):183. doi: 10.1186/s13075-015-0702-6. PMID 26189728
- [Background] Benichou C. Criteria of drug-induced liver disorders. Report of an international consensus meeting. J Hepatol. 1990 Sep;11(2):272-6. doi: 10.1016/0168-8278(90)90124-a. PMID 2254635
- [Background] Blakemore R, Story E, Helb D, Kop J, Banada P, Owens MR, Chakravorty S, Jones M, Alland D. Evaluation of the analytical performance of the Xpert MTB/RIF assay. J Clin Microbiol. 2010 Jul;48(7):2495-501. doi: 10.1128/JCM.00128-10. Epub 2010 May 26. PMID 20504986
- See also: Yazdany J, Dall'Era M. Definition and classification of lupus and lupus-related disorders. In: Wallace DJ, Hahn BH, editors. DUBOIS' lupus erythematosus and related syndromes. 8th edition. Philadelphia: Elsevier Saunders; 2013. pp. 1-7. — https://doi.org/10.1016/B978-0-323-47927-1.00002-5
- See also: Global tuberculosis report 2020: executive summary. © World Health Organisation 2020. — https://apps.who.int/iris/bitstream/handle/10665/337538/9789240016095-eng.pdf
- See also: Guidelines for the Prevention and Treatment of Opportunistic Infections in HIV- Infected Adults and Adolescents — https://clinicalinfo.hiv.gov/en/guidelines/adult-and-adolescent-opportunistic-infection/whats-new-guidelines
- See also: Moon JY, Kwon HM, Ahn EY, Park JK, Song YW, Lee EB. Efficacy of Isoniazid Chemoprophylaxis in Lupus Nephritis Patients [abstract]. Arthritis Rheumatol. 2015; 67 (suppl 10).(abstract). — https://acrabstracts.org/abstract/efficacy-of-isoniazid-chemoprophylaxis-in-lupus-nephritis-patients/
- See also: National Cancer Institute. Common terminology criteria for adverse events (CTCAE). — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/docs/CTCAE_v5_Quick_Reference_8.5x11.pdf
- See also: Ministry of Health of the Republic of Indonesia. National Guidelines for Medical Services: Tuberculosis Management. Jakarta (2020). — https://tbindonesia.or.id/wp-content/uploads/2024/02/Revised-NSP-TB-2020-2024-and-interim-plan-2025-2026_final_ttd-1.pdf

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT06618573/Prot_ICF_000.pdf